CLINICAL TRIAL: NCT01333878
Title: An Open-Label, Pilot Trial to Assess the Impact of Subcutaneous Abatacept in Rheumatoid Arthritis Assessing Inhibition of Structural Damage Determined by Low Field Extremity MRI (eMRI) and X-ray
Brief Title: Impact of Subcutaneous Abatacept in Rheumatoid Arthritis Assessing Inhibition of Structural Damage
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Orrin M Troum, M.D. and Medical Associates (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMS IM101-281
Record Dates: First submitted 2011-04-07; First posted 2011-04-12 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-Label Subcutaneous Abatacept (Experimental): Open-Label Subcutaneous Abatacept
  Interventions: Biological: Subcutaneous Abatacept

INTERVENTIONS:
Biological: Subcutaneous Abatacept — Subcutaneous Abatacept 125 mg once weekly for 6 months

SUMMARY:
The hypothesis of this study is that subcutaneous Abatacept is effective in reducing synovial inflammation, osteitis, and erosions in Rheumatoid Arthritis as assessed by low field extremity MRI and X-ray.

DETAILED DESCRIPTION:
This is an open-label study of the efficacy of subcutaneous (SC) Abatacept to inhibit progression of structural joint damage in patients with active rheumatoid arthritis (RA) receiving MTX and have inadequate disease control (defined as an ESR based DAS28 ≥ 3.2 AND ≥ 6 swollen and ≥ 6 tender joints). The study consists of a screening period (Days -21 to -7), a baseline visit (Days -20 to -1), and a treatment Period (open label Abatacept 125 mg SC for 24 weeks). All the visits may occur at the indicated week +/- 2 days. The last efficacy assessments are to be conducted at Week 24 and subjects are to be contacted by telephone for a safety follow-up 2 months after the final study agent has been administered.

The maximum length of the study is 35 weeks, which includes the 2-week screening period, 1-week baseline period, 24-week open label treatment, and 8-week follow-up period. Eligible subjects are to continue their current MTX treatment regimen, a stable dose of at least 15mg/week, during the entire length of the study (24 weeks). At Day 0, patients who meet inclusion criteria, will be dosed from Day 0 to Week 24 with Abatacept 125 mg SC injection.

Subjects are to self-administer SC study agent at Weeks 5, 6, 7, 9, 10, 11, 13, 14, 15, 17, 18, 19, 21, 22, and 23 and are not required to return to the study site at these weeks. All other visits, SC study agent is to be administered while the subject is at the study site.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects currently experiencing active moderate to severe RA according to the revised 1987 ACR criteria for the diagnosis of RA at screening. The ESR-based DAS 28 must be equal or greater than 3.2
2. MTX inadequate responders with moderate to severe RA. Subjects currently receiving MTX for at least 12 weeks and who have received MTX at a stable dose (≥15mg/week) for at least 6 weeks prior to treatment (Day 0). They must be biologic drug naive
3. All subjects must receive at least 5 mg oral folic acid weekly.
4. At screening active RA as defined by ≥ 6 swollen joints and ≥ 6 tender joints with erythrocyte sedimentation rate (ESR) ≥ 28 mm/h.
5. Subjects must be seropositive with documented rheumatoid factor (RF) or anti-cyclic citrullinated peptide (anti CCP) positivity. If a documented history of RF or anti CCP positivity is not available, RF and anti CCP titers will be obtained at screening
6. MRI evidence of at least one joint with osteitis or erosion attributable to RA as determined by an MRI musculoskeletal radiologist. Any joint of the dominant hand or wrist can be considered with the exception of distal interphalangeal joints of the hands.
7. If subjects are receiving an oral corticosteroid, the dose must be ≤10 mg/day prednisone (or equivalent) and stable for at least 28 days prior to treatment (Day 0).
8. Subjects able and willing to give written informed consent and comply with the requirements of the study protocol. Informed consent must be obtained prior to any study-related procedures.

   A copy of the signed informed consent form must be given to the subject
9. Subjects must be willing to self-inject or allow a caregiver to administer the subcutaneous injection

Exclusion Criteria:

1. Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization
2. Rheumatic autoimmune disease other than RA, including systemic lupus erythematosus (SLE), mixed connective tissue disease (MCTD), scleroderma, polymyositis, or significant systemic involvement secondary to RA (vasculitis, pulmonary fibrosis or Felty's syndrome). Prior history of or current inflammatory joint disease other than RA (gout, Lyme disease, seronegative spondyloarthropathy including reactive arthritis and psoriatic arthritis)
3. Functional class IV as defined by the ACR Classification of Functional Status in RA
4. Current treatment with any traditional DMARDs other than MTX within 4 weeks before the screening visit
5. Treatment with any investigational agent within 4 weeks (or 5 half-lives of investigational agent, whichever is longer) before screening
6. Exposure to any Biologic Response Modifying Agent
7. Intra Articular or parenteral corticosteroids within 6 weeks prior to screening
8. Immunization with live vaccine within 3 months prior to enrollment and a need for a live vaccine during the study
9. Subjects who have a metal device where the use of MRI is contraindicated (e.g.,any type of electronic, mechanical, or magnetic implant; cardiac pacemaker, aneurysm clip; implanted cardioverter defibrillator; or a cochlear implant). Subjects who have a potential ferromagnetic foreign body (metal shavings, metal slivers, other metal objects) for which they have sought medical attention
10. Exclusionary laboratory: Serum creatinine >2 mg/dL, ALT or AST > 2.0 x ULN, total bilirubin > 2.0 x ULN, platelet count <100 x 109 /L, hemoglobin < 8.5 g/dL, WBC count < 1,000/mm3 , absolute neutrophil count < 1,000/ mm3, absolute lymphocyte count < 500/mm3, positive HBsAg or HCV antibody, or positive HIV test.
11. Pregnant women or nursing mothers
12. Females of child bearing potential who are not using reliable means of contraception
13. Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary, renal, hepatic, endocrine or GI disease
14. Uncontrolled disease states, such as asthma, psoriasis, or inflammatory bowel syndrome, where flares are commonly treated with corticosteroids
15. Known active current or history of recurrent bacterial, viral, fungal, mycobacterial, or other infections such as atypical mycobacterial disease, hepatitis B and C, HIV, herpes zoster, or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening.
16. A history of active TB within the last 3 years even if it was treated. A history of active TB greater than 3 years ago unless there is documentation that the prior anti-TB treatment was appropriate in duration and type. A positive PPD skin test (≥5 mm) or positive QuantiFERON-TB Gold serum test without appropriate prophylaxis (at least 1 month of the planned local guidelines treatment regimen)
17. Any malignancy except for skin cancer (basal cell or squamous cell) diagnosed within the previous 5 years
18. History of alcohol, drug, or chemical abuse
19. Neuropathies or other painful conditions that might interfere with pain evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-03; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Inhibition & progression of structural damage | 6 months
  Assess inhibition & progression of structural damage in MTX inadequate responders with moderate to severe active RA on SC Abatacept plus MTX, utilizing eMRI and X-ray at baseline, eMRI at Week 12, and eMRI and X-ray final assessment at week 24.

SECONDARY OUTCOMES:
Improvement in ESR-based DAS28 | 6 months
  Assess improvement in ESR-based DAS28, physician global assessment, and improvement in HAQ score

CONTACTS AND LOCATIONS:
Overall Officials: Orrin M Troum, MD, Principal Investigator — Orrin M. Troum, MD & Medical Associates
Locations (1):
- Orrin M. Troum, MD and Medical Associates, Santa Monica, California, United States